CLINICAL TRIAL: NCT05265481
Title: The Effect of Tapping in the Venous Dilatation for Peripheral IV Access
Acronym: Tapping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB202102042
Record Dates: First submitted 2022-01-31; First posted 2022-03-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Catheterization, Peripheral; Venous Dilatation
Keywords: Catheterization, Peripheral; Massaging; Tapping; Tourniquet; Venipuncture; Venodilation
MeSH Terms: interventions — Tourniquets

STUDY DESIGN:
Intervention Model Description: The investigators will make the measurements four times for each vein and participant:
  1. Baseline: In this phase, the investigators will not apply any venodilation method
  2. Tourniquet applied: The investigators will apply a blood pressure cuff tourniquet inflated to 60 mmHg pressure.
  3. Tourniquet plus tapping directly over the vein manually
  4. Tourniquet plus tapping directly over the vein with a massage device The investigators will change the 3rd and 4th items between two arms of the same participant. In other words, the investigators will do 1-2-3-4 for a left arm but 1-2-4-3 for the right arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baseline (No Intervention): In this phase, the investigators will not apply any venodilation method.
- Tourniquet applied (Active Comparator): The investigators will apply a blood pressure cuff tourniquet inflated to 60 mmHg pressure.
  Interventions: Device: Tourniquet
- Tourniquet plus manual tapping (Active Comparator): The investigators will apply a pressure cuff tourniquet inflated to 60 mmHg plus tapping directly over the vein manually.
  Interventions: Device: Tourniquet; Device: Manual Tapping
- Tourniquet plus device tapping (Experimental): The investigators will apply a pressure cuff tourniquet inflated to 60 mmHg plus tapping directly over the vein with a massage device.
  Interventions: Device: Tourniquet; Device: Device tapping

INTERVENTIONS:
Device: Tourniquet — The investigators will apply a pressure cuff tourniquet inflated to 60 mmHg
  Arms: Tourniquet applied; Tourniquet plus device tapping; Tourniquet plus manual tapping
Device: Manual Tapping — The investigators will apply tapping directly over the vein manually to increase the vein dimension.
  Arms: Tourniquet plus manual tapping
Device: Device tapping — The investigators will apply tapping directly over the vein with a massage device to increase the vein dimension.
  Arms: Tourniquet plus device tapping

SUMMARY:
Peripheral intravenous cannulation (PIVC) is one of the most common interventions in medical practice. Venous dilatation is helpful for successful PIV placement. Several techniques include hot pack application, tourniquet, massaging, and tapping over the vein to increase vein caliber described in the literature. However, none of them has been rigorously studied. Therefore, there is still no 'best practice' on how to effect vein dilation in a standard way.

This study aims to investigate the effect of standardized tapping on venous dilatation with a massage device compared to manual non-standardized tapping and define a standard tapping technique using a device.

In this study, the investigators also aim to investigate the effect of tourniquet application with and without vein tapping effect on peripheral vein caliber as determined by ultrasound measurement.

DETAILED DESCRIPTION:
PIVC is one of the most common medical interventions in daily practice. Even though it seems like it should be an easy procedure, PIVC can be challenging.

Venous dilatation optimizes conditions for successful vein cannulation. Several techniques are described to affect venodilation, but none of them are standardized because they are done manually, and there will be individual variations among clinicians.

Tapping over the vein has been reported as an effective method. It has been hypothesized that tapping affects vein vaso-nervorum activation and local histamine release. Tapping or massage over the cannulation site is readily applied in busy medical practice, with a third of nurses using tapping or massage to promote venodilation. Tapping and massage are effective methods of vasodilatation to make the vein more prominent for venipuncture, with tapping more effective than massage (Ichimura et al.) There are limited data concerning the effect of tapping in PIVC and its standardization. In the current literature, there is no standard technique on how tapping should be performed.

Specific Aims:

* H0: Standardized tapping with a massage device is not an effective technique to dilate the peripheral veins for PIVC compared to manual tapping.
* H1: Standardized tapping with a device is a more effective technique to dilate peripheral veins for PIVC compared to manual tapping.

The investigators expect to learn to what degree a tourniquet increases peripheral vein size and to what degree that is augmented by tapping.

Research Plan:

This is a prospective non-randomized, controlled, non-invasive intervention study.

The investigators will visually and also with surface ultrasound inspect the upper extremity. The investigators will not get blood tests or X-rays for study purposes. The investigators will measure the venous diameter of a vein or veins on the back of the hand and deeper within the forearm and in the antecubital fossa using ultrasound. The investigators will use a survey including participant's demographics (age, gender, handedness, smoking history)

The investigators will use a portable ultrasound device (Butterfly iQ+, Butterfly Network, Inc., CT, USA) connected to an iPad to record ultrasound images (as pictures) and measure the diameter and cross-section area of the various veins. The investigators will take vein measurements from the dorsal hand, cubital, and mid-forearm regions. The investigators will take the measurements from the midline of the antecubital, volar side of the forearm, and dorsal hand regions. The investigators will put masking tapes on the skin as a reference point to make all the measurements from the same plane."

Then the investigators will determine the midpoint of the forearm, the antecubital site, and the volar wrist crease. The midpoint of this line will be the mid-forearm vein measurement site. The investigators will use superficial dorsal hand veins of the dorsal metacarpal region for the dorsal hand vein measurements. During the baseline measurements, the investigators will get the best image with ultrasound and then mark the skin to get all the measurements from the same cross-sectional area and place water-resistant tape with a scale.

The investigators will not use ultrasound gel or direct ultrasound probe application to the skin to prevent any possible ultrasound transducer-related venous compression. Instead, the investigators will sufficiently submerge the hand, forearm, and elbow in a fresh room temperature water-filled basin to allow precise vein caliber measurements with an ultrasound probe without any probe contact with the skin. This technique provides high-quality ultrasound images of superficial and deep veins.

The investigators will use a standard adult blood pressure cuff applied to the mid-upper arm statically inflated to 60mmHg to serve as a tourniquet.

The investigators will measure these parameters:

* AP diameter of the vein
* The cross-sectional area of the vein
* Width of the vein The investigators will measure veins from three different locations
* Anterior antecubital superficial vein
* Volar mid-forearm region deep vein
* Dorsal hand superficial vein

The investigators will make the measurements four times for each vein and participant:

1. Baseline: In this phase, the investigators will not apply any venodilation method
2. Tourniquet applied: The investigators will apply a blood pressure cuff tourniquet inflated to 60 mmHg pressure.
3. Tourniquet plus tapping directly over the vein manually
4. Tourniquet plus tapping directly over the vein with a massage device The investigators will change the 3rd and 4th items between two arms of the same participant. In other words, the investigators will do 1-2-3-4 for a left arm but 1-2-4-3 for the right arm. The investigators will assess whether the order affects the vein diameter by this change. The venous blood pressure cuff tourniquet will not be applied for more than 20 minutes continuously.

The investigators will take photos of the ultrasound vein visualizations and measure the diameter and cross-sectional area. This will have no PHI attached to the ultrasound images.

The investigators will take photos of the skin using a calibration ruler to assess the dilation of the visible veins externally. These photos will not reveal the subject's face or any personally identifiable images or information. After all study procedures are complete on the initial arm, study procedures will be repeated on the opposite arm.

Primary investigators will be responsible for collecting the data.

The investigators will not use the name or identifiable data when entering the data into the software. Rather than that, the investigators will code the participants (E.g., A01, B02). This data will be stored only in the departmental password-protected encrypted share drive. The survey and paperwork, including any participant data, will be stored at the locked drawers in investigators' offices

ELIGIBILITY:
Inclusion Criteria:

* >18 years old,
* Giving informed consent,
* COVID-19 vaccinated (proof of vaccination must be shown)

Exclusion Criteria:

* COVID-19 unvaccinated,
* Having unexplained COVID symptom(s) (This will be assessed by asking the ONE.UF screening questions):

  * Fever or chills
  * Cough
  * Fatigue
  * Muscle or body aches
  * Headache
  * New loss of taste or smell
  * Sore throat
  * Congestion or runny nose
  * Nausea or vomiting
  * Diarrhea
  * Close contact with a COVID-19 patient in 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-07 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in standardized tapping with a device for PIVC | 2 hours
  The primary outcome is to measure the vein diameters after manual and device tapping and detect the change from baseline in vein diameters.

SECONDARY OUTCOMES:
Change in the effect of tourniquet application | 2 hours
  Secondary outcome is to measure the vein diameters before and after tourniquet application and detect the change from baseline in vein diameters.

CONTACTS AND LOCATIONS:
Overall Officials: Brandi Lattinville, Study Director — University of Florida; Yahya A Acar, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There will be no Data Safety Monitoring Board (DSMB) or an oversight committee for the study and no individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Yasuda K, Sato S, Okada K, Yano R. The venodilation effects of tapping versus massaging for venipuncture. Jpn J Nurs Sci. 2019 Oct;16(4):491-499. doi: 10.1111/jjns.12261. Epub 2019 Jun 20. PMID 31222981
- [Background] Ichimura M, Matsumura Y, Sasaki S, Murakami N, Mori M, Ogino T. The characteristics of healthy adults with hardly palpable vein--Relations between easy venous palpation and physical factors. Int J Nurs Pract. 2015 Dec;21(6):805-12. doi: 10.1111/ijn.12313. Epub 2014 Apr 14. PMID 24724700
- [Background] Ichimura M, Sasaki S, Mori M, Ogino T. Tapping but not massage enhances vasodilation and improves venous palpation of cutaneous veins. Acta Med Okayama. 2015;69(2):79-85. doi: 10.18926/AMO/53336. PMID 25899629